CLINICAL TRIAL: NCT06298344
Title: The Role of Thiamine on Left Ventricular Structure and Function After Transcatheter Closure Through the Examination of MMP-9 Dan TIMP-1 in Children With Left-to-Right Shunt Congenital Heart Disease
Brief Title: The Role of Thiamine After Transcatheter Closure in Children With Left-to-Right Shunt Congenital Heart Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Putri Amelia, dr. Putri Amelia, M.Ked (Ped), Sp.A(K), Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2024-02-21; First posted 2024-03-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Congenital Heart Disease; Thiamine Deficiency; Patent Ductus Arteriosus; Ventricular Septal Defect; Atrial Septal Defect
MeSH Terms: conditions — Heart Defects, Congenital; Thiamine Deficiency; Ductus Arteriosus, Patent; Heart Septal Defects, Ventricular; Heart Septal Defects, Atrial | interventions — Thiamine

STUDY DESIGN:
Intervention Model Description: Double blind
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thiamine (Experimental): Patients with left to right shunt congenital heart disease who undergone transcatheter closure Intervention: Daily Thiamine 100 mg in 28 days.
  Interventions: Drug: Thiamine
- Placebo (No Intervention): Patients with left to right shunt congenital heart disease who undergone transcatheter closure Interventions: Daily Placebo oral (Manufactured to mimic Thiamine) in 28 days.

INTERVENTIONS:
Drug: Thiamine — Daily Thiamine 100 mg in 28 days
  Other Names: Vitamin B1
  Arms: Thiamine

SUMMARY:
Currently, research on the effect of thiamine administration during transcatheter closure on the structure and function of the left ventricle by examining levels of matrix metalloproteinase-9 and tissue inhibitor of metalloproteinase-1 in children with left to right shunt congenital heart disease has never been carried out in Indonesia, so it is necessary carried out this research. This research was carried out by administering 100 mg of thiamine once per day to patients post transcatheter closure for 28 days. The parameters assessed were MMP-9, TIMP-1, and echocardiography to assess the structure and function of the left ventricle in CHD patients with left to right shunt lesions.

DETAILED DESCRIPTION:
Specifically the investigators want to study about :

1. The differences in serum levels of matrix metalloproteinase-9 in patients with congenital heart disease with left to right shunt lesions after transcatheter closure who received thiamine and those who did not receive thiamine.
2. The differences in serum tissue inhibitor of metalloproteinase-1 levels in patients with congenital heart disease with left to right shunt lesions after transcatheter closure who received thiamine and those who did not receive thiamine.
3. The differences in left ventricular structure in patients with congenital heart disease with left to right shunt lesions after transcatheter closure who receive thiamine and those who do not receive thiamine.
4. The differences in left ventricular function in patients with congenital heart disease with left to right shunt lesions after transcatheter closure who receive thiamine and those who do not receive thiamine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 6 months - 18 years.
2. Patients diagnosed with left to right shunt lesion CHD with heart failure based on ROSS or NYHA criteria.
3. Patients who will undergo intervention with transcatheter closure.

Exclusion Criteria:

1. Patients who experienced acute infections before the procedure.
2. There are other heart defects that require surgery.
3. There is a hereditary, genetic disorder, syndrome or other chronic disease.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between transcatheter closure and left ventricular structure change after thiamine treatment | 1 day before transcather closure and 28 days after trancatheter closure
  The left ventricular structure of each participant is measured with echocardiography at the beginning and the end of the study and then the investigators calculate the left ventricular structure change (in percentage, %)

SECONDARY OUTCOMES:
Correlation between transcatheter closure and left ventricular function change after thiamine treatment | 1 day before transcather closure and 28 days after trancatheter closure
  The left ventricular function of each participant is measured with echocardiography at the beginning and the end of the study and then the investigators calculate the left ventricular function change (in percentage, %)
Correlation between transcatheter closure and serum matrix metalloproteinase-9 level change after thiamine treatment | 1 day before transcather closure and 28 days after trancatheter closure
  The serum matrix metalloproteinase-9 level of each participant is measured at the beginning and the end of the study and then the investigators calculate the level change (in percentage, %)
Correlation between transcatheter closure and serum tissue inhibitor of metalloproteinase-1 level change after thiamine treatment | 1 day before transcather closure and 28 days after trancatheter closure
  The serum tissue inhibitor of metalloproteinase-1 level of each participant is measured at the beginning and the end of the study and then the investigators calculate the level change (in percentage, %)

CONTACTS AND LOCATIONS:
Overall Officials: Putri Amelia, Principal Investigator — Universitas Sumatera Utara
Locations (1):
- RSUP H Adam Malik, Medan, North Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No